CLINICAL TRIAL: NCT02992938
Title: Administration of Acetazolamide to Prevent Remifentanil Induced Hyperalgesia: Randomize Double Blind Clinical Trial
Brief Title: Administration of Acetazolamide to Prevent Remifentanil Induced Hyperalgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Gutiérrez, MD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 803/16
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Hyperalgesia; Opioid-Related Disorders
Keywords: Opioid hyperalgesia; Acetazolamide; Remifentanil
MeSH Terms: conditions — Hyperalgesia; Opioid-Related Disorders | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetazolamide (Experimental): 250 mg VO of acetazolamide will be administered the day of the surgery 2 hours before anesthesia induction
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): An oral tablet without active principle acetazolamide but with the same physical characteristics will be administered the day of the surgery 2 hours before anesthesia induction
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Acetazolamide
Drug: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
Remifentanil is a potent opioid widely used during the administration of general anesthesia. There is a lot of evidence that suggest that the used of remifentanil is associated with the development of hyperalgesia (a reduction of nociceptive thresholds). However, the mechanism of this hyperalgesia is not fully understood.

Recently, it was demonstrated that the disruption of the Cl- homeostasis could be involved. Interestingly, this was prevented in a murine model with the administration of Acetazolamide, a carbonic anhydrase inhibitor. In our clinical trial we will try to determine if the preoperative administration of acetazolamide could prevent the hyperalgesia induced by remifentanil in patients scheduled for thyroidectomy with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thyroidectomy with general anesthesia in the University of Chile Clinical Hospital

Exclusion Criteria:

* Patients ASA III y IV
* Chronic pain history
* Drug and alcohol abuse
* Chronic use of opioid and sedatives
* Neuropsychiatric illness
* NSAID and other analgesics used the 48 hours previous to the surgery
* CMI > 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Change in the mechanical pain threshold in an area distant to the site of the injury | 12-18 hours after the end of the surgery
  The threshold will be determine using von Frey monofilaments before the surgery and will be compared 12-18 hours after the end of the surgery

SECONDARY OUTCOMES:
Change in the mechanical pain threshold in an area distant to the site of the injury | 2 hours after the end of the surgery
Postoperative pain | The first postoperative day
  A visual analogue scale (VAS; 0, no pain; 100, worst poss- ible pain) will be used to assess pain
Morphine consumption | The first postoperative day
  Morphine consumption with a patient controlled analgesia (PCA) in mg

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Gutierrez, MD, Principal Investigator — Anesthesia Department, University of Chile; Antonello Penna, MD PhD, Principal Investigator — Anesthesia Department, University of Chile
Locations (1):
- Faculty of Medicine, University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferrini F, Trang T, Mattioli TA, Laffray S, Del'Guidice T, Lorenzo LE, Castonguay A, Doyon N, Zhang W, Godin AG, Mohr D, Beggs S, Vandal K, Beaulieu JM, Cahill CM, Salter MW, De Koninck Y. Morphine hyperalgesia gated through microglia-mediated disruption of neuronal Cl(-) homeostasis. Nat Neurosci. 2013 Feb;16(2):183-92. doi: 10.1038/nn.3295. Epub 2013 Jan 6. PMID 23292683
- [Result] Echevarria G, Elgueta F, Fierro C, Bugedo D, Faba G, Iniguez-Cuadra R, Munoz HR, Cortinez LI. Nitrous oxide (N(2)O) reduces postoperative opioid-induced hyperalgesia after remifentanil-propofol anaesthesia in humans. Br J Anaesth. 2011 Dec;107(6):959-65. doi: 10.1093/bja/aer323. Epub 2011 Sep 28. PMID 21965050
- [Result] Angst MS, Koppert W, Pahl I, Clark DJ, Schmelz M. Short-term infusion of the mu-opioid agonist remifentanil in humans causes hyperalgesia during withdrawal. Pain. 2003 Nov;106(1-2):49-57. doi: 10.1016/s0304-3959(03)00276-8. PMID 14581110
- [Result] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467